CLINICAL TRIAL: NCT02312726
Title: Postplacental Intrauterine Device Insertion: A Mixed Methods Assessment of Women's Experience
Acronym: PIPPI
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Other Study IDs: UNM HSC 13-440
Record Dates: First submitted 2014-10-23; First posted 2014-12-09 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Contraception
Keywords: mixed methods; visual analog scale; verbal rating score; pain assessment; patient satisfaction; contraceptive devices; postpartum
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Epidural group: Participants who elect to have an epidural anesthesia during labor, delivery and postplacental IUD insertion
  Interventions: Procedure: Postplacental IUD insertion
- Non Epidural group: Participants who elect not to have epidural anesthesia during labor, delivery and postplacental IUD insertion
  Interventions: Procedure: Postplacental IUD insertion

INTERVENTIONS:
Procedure: Postplacental IUD insertion — Postplacental IUD insertion using the standardized ring forceps technique (Speroff and Mishell 2008) under ultrasound guidance, within 10-30 minutes of vaginal delivery.
  Other Names: Immediate postpartum IUD insertion

SUMMARY:
The primary objective of this mixed methods pilot study is to understand women's experiences with postplacental intrauterine device (IUD) insertion through postpartum semi-structured interviews. For secondary objectives, the investigators will collect visual analog scale (VAS) and verbal rating score (VRS) data on women's pain experienced just before and immediately after IUD insertion. The investigators will perform postpartum interviews in each group until we reach thematic saturation. The investigators will recruit at least 60 women (30 each in the epidural and no epidural group) from the University of New Mexico Hospital (UNMH) affiliated antenatal clinics to conduct our quantitative data analysis.

DETAILED DESCRIPTION:
Postplacental IUD insertion following vaginal or cesarean delivery is as effective in preventing pregnancy as interval insertion, and it is utilized more often in other countries such as China, Mexico and Egypt compared with the US (Celen, Moroy et al. 2004; Eroglu, Akkuzu et al. 2006; Kapp and Curtis 2009; Grimes, Lopez et al. 2010). In addition, current evidence supports the safety and superior cost effectiveness of IUD use (Trussell, Lalla et al. 2009; ACOG 2011). Postplacental IUD insertion is practiced routinely in US hospitals with active family planning faculty (including University of New Mexico Hospital), and has become standard of care for postpartum contraception options counseling in these institutions. Despite ample evidence supporting the safety and effectiveness of postplacental IUD insertion, the practice is uncommon among US providers and many women remain unaware of this option. Reasons for underutilization in the US may include lack of reimbursement, sufficient provider knowledge and training, and patient awareness.

Postplacental IUD insertion is also an attractive method for provision of postpartum contraception for several reasons: women are motivated to initiate contraception, they are not pregnant, and access to medical care is readily available.

Pain is a subjectively complex and universal experience which encompasses more experiential aspects than objective measurements of physical pain can capture. We know that interval IUD placement is painful, and that anxiety and fear of pain can be a barrier to IUD uptake, particularly among adolescent women (Allen, Bartz et al. 2009). Pain and low satisfaction with the IUD insertion procedure may limit patients' endorsement of the method to other women. There is insufficient research examining the patient's subjective experience with postplacental IUD placement. In addition, there is limited data about the physical pain level associated with postplacental IUD insertion.

Several studies have examined the efficacy of interventions to reduce pain for interval IUD insertion for nulliparous and multiparous women (Hubacher, Reyes et al. 2006; Edelman, Schaefer et al. 2011; Maguire, Davis et al. 2012; Swenson, Turok et al. 2012). Procedural aspects and clinical circumstances of postplacental IUD insertion differ substantially from those associated with interval insertion, preventing extrapolation of findings from studies of interval IUD insertion to postplacental insertion.

Specific aims:

1. Obtain an understanding of women's experiences with ring forceps postplacental IUD insertion through semi-structured interviews conducted prior to discharge from the hospital.
2. Establish objective assessments of physical pain associated with ring forceps postplacental IUD insertion using the 100mm Visual Analog Scale (VAS) and a categorical Verbal Rating Scale (VRS).

Participants will be recruited within the third trimester of pregnancy, when standard counseling typically occurs to address postpartum contraception options with patients; this usually occurs at 30 weeks gestation or later. The pain score assessment and interview data collection for each participant will take place while the patient is admitted for vaginal delivery at the University of New Mexico Hospital (UNMH).

The primary and secondary endpoints will occur at the conclusion of study enrollment when the last postpartum interview has been completed (when we have reached thematic saturation), and when we have at least 30 pain score assessments for the epidural and no epidural groups. The study is not designed to detect a difference in VAS scores between those women who have an epidural and those who do not (a power analysis was not performed), but rather this secondary objective is intended to establish the mean VAS score for each group. Because women will not know for certain if they will elect a labor epidural at the time of antenatal recruitment and because some women may not get undergo postplacental IUD placement for obstetric reasons (e.g., chorioamnionitis, postpartum bleeding, etc), it may be necessary to recruit more women than needed to achieve 30 women for each group. Up to 175 women will be recruited in the study.

When a participant presents to UNMH L&D to deliver her baby, we will confirm her ongoing desire to participate in the study, and will review the expectations for participation. We will confirm that the subject continues to meet the inclusion and exclusion criteria. Following vaginal birth, all eligible participants will undergo postplacental IUD insertion using the standardized ring forceps technique under ultrasound guidance, within 10-30 minutes of vaginal delivery, per standard of care for this procedure.

We will obtain a VAS and VRS score after the placenta delivers and prior to inserting the IUD, and a second set of scores within 5 minutes of insertion. We will assess provider ease of procedure using a four-point Likert scale. Prior to discharge from the hospital, we will confirm that subjects remain willing to participate in the postpartum interview portion of the study. If they elect to continue participation, they will undergo a semi-structured interview designed to explore their perceptions of the postpartum IUD insertion experience. Participants will have an appointment with their primary obstetric providers within two weeks of delivery for an IUD string check, per standard of care. We will not collect data from the postpartum IUD string check visit.

Data will be managed with the following methods: 1) Only the research team will have access to the data; 2) The data will be stored separately from consents; 3) Data sheets will be coded with the participant's assigned study code.

Data will be stored using the following methods: 1) The UNM Redcap database reposing study data will not contain unique patient identifiers; 2) The database for both quantitative and qualitative data will be stored on a secure, password protected server; 3) The identifiers will be linked to the patient's code number on a spreadsheet in a secure, designated password protected computer in the UNMH Ob-Gyn Department.

Data will be destroyed using the following methods: 1) Audio recordings of the interviews will be erased once they have been transcribed; 2) The link between study code and unique participant identifiers will be destroyed when the study is closed through the UNM Human Research Protections Office; 3) Study records will be kept for a minimum of three years; 4) HIPAA authorizations will be retained for a minimum of six years.

This study poses not more than minimal risk to subjects. There is a small risk that protected health information will be identified with study data. Study participation may be considered inconvenient by subjects.

The subjects will be permitted to withdraw from the study at any time without any effect on their access or options for care. The investigators have the right to end a subject's participation in this study if they determine that she no longer meets inclusion or exclusion criteria or if they, for whatever reason, believe that it is not in her best interests to continue participation. The investigators may also withdraw a subject if they determine that the subject is not following study protocol.

No further data collection will occur on a participant who withdraws from this study. The Institutional Review Board (IRB) will be notified of such withdrawals per IRB protocol.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking or Spanish-speaking only (SSO) women
* Women who express a desire to have an IUD inserted immediately following anticipated vaginal delivery.

Exclusion Criteria:

* Unanticipated cesarean delivery
* Chorioamnionitis
* Significant postpartum hemorrhage (estimated blood loss requiring intervention beyond standard therapy and not resolved within approximately 10 minutes)
* Third or fourth degree obstetric vaginal laceration
* Manual extraction of the placenta
* Untreated gonorrhea, chlamydia and/or trichomoniasis
* Known or suspected distorted uterine cavity
* Current use of controlled substances for chronic pain management
* Current substance abuse/ addiction.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit women from the University of New Mexico Hospital (UNMH) affiliated antenatal clinics. We will also recruit women from the UNMH obstetric units, provided the women are not in labor. Women will be approached about participation in the study if, after routine antenatal contraceptive counseling conducted in the third trimester, they report that they would like to undergo postplacental IUD insertion. We will use convenience sampling.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rameet H Singh, MD, MPH, Principal Investigator — UNM OB GYN Division of Family Planning
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] ACOG Practice Bulletin No. 121: Long-acting reversible contraception: Implants and intrauterine devices. Obstet Gynecol. 2011 Jul;118(1):184-196. doi: 10.1097/AOG.0b013e318227f05e. No abstract available. PMID 21691183
- [Background] Allen RH, Bartz D, Grimes DA, Hubacher D, O'Brien P. Interventions for pain with intrauterine device insertion. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD007373. doi: 10.1002/14651858.CD007373.pub2. PMID 19588429
- [Background] Celen S, Moroy P, Sucak A, Aktulay A, Danisman N. Clinical outcomes of early postplacental insertion of intrauterine contraceptive devices. Contraception. 2004 Apr;69(4):279-82. doi: 10.1016/j.contraception.2003.12.004. PMID 15033401
- [Background] Edelman AB, Schaefer E, Olson A, Van Houten L, Bednarek P, Leclair C, Jensen JT. Effects of prophylactic misoprostol administration prior to intrauterine device insertion in nulliparous women. Contraception. 2011 Sep;84(3):234-9. doi: 10.1016/j.contraception.2011.01.016. Epub 2011 Mar 3. PMID 21843686
- [Background] Eroglu K, Akkuzu G, Vural G, Dilbaz B, Akin A, Taskin L, Haberal A. Comparison of efficacy and complications of IUD insertion in immediate postplacental/early postpartum period with interval period: 1 year follow-up. Contraception. 2006 Nov;74(5):376-81. doi: 10.1016/j.contraception.2006.07.003. Epub 2006 Sep 15. PMID 17046378
- [Background] Grimes DA, Lopez LM, Schulz KF, Van Vliet HA, Stanwood NL. Immediate post-partum insertion of intrauterine devices. Cochrane Database Syst Rev. 2010 May 12;(5):CD003036. doi: 10.1002/14651858.CD003036.pub2. PMID 20464722
- [Background] Hubacher D, Reyes V, Lillo S, Zepeda A, Chen PL, Croxatto H. Pain from copper intrauterine device insertion: randomized trial of prophylactic ibuprofen. Am J Obstet Gynecol. 2006 Nov;195(5):1272-7. doi: 10.1016/j.ajog.2006.08.022. PMID 17074548
- [Background] Kapp N, Curtis KM. Intrauterine device insertion during the postpartum period: a systematic review. Contraception. 2009 Oct;80(4):327-36. doi: 10.1016/j.contraception.2009.03.024. Epub 2009 Aug 29. PMID 19751855
- [Background] Maguire K, Davis A, Rosario Tejeda L, Westhoff C. Intracervical lidocaine gel for intrauterine device insertion: a randomized controlled trial. Contraception. 2012 Sep;86(3):214-9. doi: 10.1016/j.contraception.2012.01.005. Epub 2012 Feb 9. PMID 22325115
- [Background] Speroff L, Mishell DR Jr. The postpartum visit: it's time for a change in order to optimally initiate contraception. Contraception. 2008 Aug;78(2):90-8. doi: 10.1016/j.contraception.2008.04.005. Epub 2008 Jun 12. No abstract available. PMID 18672108
- [Background] Swenson C, Turok DK, Ward K, Jacobson JC, Dermish A. Self-administered misoprostol or placebo before intrauterine device insertion in nulliparous women: a randomized controlled trial. Obstet Gynecol. 2012 Aug;120(2 Pt 1):341-7. doi: 10.1097/AOG.0b013e31825d9ec9. PMID 22825094
- [Background] Trussell J, Lalla AM, Doan QV, Reyes E, Pinto L, Gricar J. Cost effectiveness of contraceptives in the United States. Contraception. 2009 Jan;79(1):5-14. doi: 10.1016/j.contraception.2008.08.003. Epub 2008 Sep 25. PMID 19041435

RESULTS

PARTICIPANT FLOW:
Groups:
- Excluded: Participants who did not meet inclusion criteria or declined after consent.
Period: Overall Study
Arm/Group | Epidural Group | Non Epidural Group | Excluded
Started | 38 | 30 | 67
Completed | 38 | 30 | 0
Not Completed | 0 | 0 | 67

BASELINE CHARACTERISTICS:
Groups:
- Total Participants Enrolled in Study: Participant characteristics for those enrolled in the study, in both the epidural and non-epidural group
Arm/Group | Total Participants Enrolled in Study
Number analyzed (Participants) | 68
Age, Customized [Median (Full Range); unit: years]
  Median Age | 27 [18 to 43]
Sex/Gender, Customized [Number; unit: participants]
  Female | 68
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 61
  African American | 1
  American Indian/Alaskan | 4
  Asian American | 1
  White | 1
Region of Enrollment [Number; unit: participants]
  United States | 68
Education [Number; unit: participants]
  Did not complete high school | 21
  Completed high school/ GED | 28
  In college/completed some college | 16
  Completed college | 3
Employment [Number; unit: participants]
  Employed part time | 8
  Employed full time | 8
  Student | 7
  Homemaker | 31
  Temporary work leave | 2
  Unemployed | 12
Income [Number; unit: participants]
  Less than $20,000 | 39
  $20,000 - $40,000 | 23
  $40,000 - $60,000 | 3
  $60,000 - $80,000 | 1
  Declined to answer | 2
Language of Preference [Number; unit: participants]
  English | 38
  Spanish | 30
Insurance [Number; unit: participants]
  None | 39
  Medicaid | 26
  Commercial | 3

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Women's Experiences With Ring Forceps Postplacental IUD Placement Through Semi-structured Interviews
Description: A semi-structured interview guide(available in both English and Spanish) which was developed in consultation with an expert in qualitative methodology at the UNM Clinical & Translational Science Center (CTSC), and UNMH family planning experts, will be administered to all participants. The interview will incorporate the following domains of women's perceptions of the postplacental IUD insertion experience: decisional influence, experience during the procedure, decisional regret, prior knowledge/ awareness of the method and postpartum contraception in general. The interview will conclude with an overall patient satisfaction score measured on a five-point Likert scale: 1 = very dissatisfied, 2 = somewhat dissatisfied, 3 = neutral, 4 = somewhat satisfied, 5 = very satisfied.
Time Frame: Within 24-48 hours after vaginal delivery, prior to hospital discharge
Population: 21 participants (out of the 68 included in the study) consented to an interview regarding their experience. We conducted 21 interviews; 9 with women who did not have an epidural and 12 with women who had an epidural.
Measure: Number; unit: participants
Arm/Group | Epidural Group | Non Epidural Group
Number analyzed (Participants) | 12 | 9
participants
  Very Satified | 12 | 7
  Satisfied | 0 | 2
  Neutral | 0 | 0
  Dissatisfied | 0 | 0
  Very Dissatisfied | 0 | 0

2. Secondary Outcome: Pain Score: Visual Analog Scale (VAS)
Description: This is a validated instrument used extensively in the assessment of acute pain. When prompted, patients will be asked to mark the continuous 100 mm VAS line at the point which most accurately represents their pain level; 0 = no pain, 100 = pain as bad as it could be.
Time Frame: Immediately prior to and within 5 minutes after IUD insertion following vaginal delivery; women who undergo a postpartum interview will be asked to perform a recall VAS pain assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Group | Non Epidural Group
Number analyzed (Participants) | 38 | 30
units on a scale
  Pre-insertion | 10.6 (15.9) | 35.3 (29.3)
  Procedure | 10.9 (19.5) | 41.4 (34.1)
  Recall | 5.4 (7.4) | 28.6 (33.2)

3. Secondary Outcome: Pain Score: Verbal Rating Scale (VRS)
Description: This is a 4-item ordinal pain scale which has been used for pain level assessment. When prompted, patients will be asked to indicate which level of pain most accurately represents their pain level; 0 = No pain, 1 = Mild pain, 2 = Moderate pain, 3 = Severe pain.
Time Frame: Immediately prior to and within 5 minutes after IUD insertion following vaginal delivery. Women who undergo a postpartum interview will be asked to perform a recal VRS pain assessment
Measure: Number; unit: participants
Arm/Group | Epidural Group | Non Epidural Group
Number analyzed (Participants) | 38 | 30
participants
  No Pain or Mild Pain before IUD placement | 34 | 15
  No Pain or Mild Pain during IUD placement | 32 | 16
  No Pain or Mild Pain at recall | 12 | 6
  Moderate Pain or Severe Pain before IUD placement | 2 | 15
  Moderate Pain or Severe Pain during IUD placement | 4 | 14
  Moderate Pain or Severe Pain at recall | 0 | 3

4. Other Pre Specified Outcome: Provider Ease-of-insertion
Description: The provider who inserts the IUD will be asked to complete a 4-item Likert scale rating perceived difficultly of insertion: 1 = easy; 2 = somewhat easy; 3 = somewhat difficult, 4 = difficult.
Time Frame: Within 5 minutes following postpartum IUD insertion
Measure: Number; unit: participants
Arm/Group | Epidural Group | Non Epidural Group
Number analyzed (Participants) | 38 | 30
participants
  Easy | 19 | 15
  Somewhat easy | 16 | 11
  Somewhat difficult | 3 | 3
  Difficult | 0 | 0
  Unanswered | 0 | 1

ADVERSE EVENTS:
Arm/Group | Epidural Group | Non Epidural Group
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/30
Other Adverse Events (participants affected / at risk) | 0/38 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No